CLINICAL TRIAL: NCT03987815
Title: Neoadjuvant Nivolumab for Operable Esophageal Squamous Cell Carcinoma
Brief Title: Neoadjuvant Nivolumab for Operable Esophageal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-01-147-0004
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2019-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): Nivolumab 240 mg fixed dose every 2 weeks, for maximum of 3 cycles
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab

SUMMARY:
This is a single arm phase II study, in which maximum 3 cycles of nivolumab (240 mg fixed dose every 2 weeks) is administered for T2- or T3-node negative esophageal squamous cell carcinoma, before curative operation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed esophageal squamous cell carcinoma
2. Clinical stage T2N0 (invasion to muscularis propria) or T3N0 (invasion to adventitia)
3. ECOG performance 0 or 1
4. Age 19 years or older

Exclusion Criteria:

1. Prior therapy (operation, radiotherapy, immunotherapy, or chemotherapy) for esophageal cancer
2. Ineligibility or contraindication for esophagectomy
3. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
4. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
5. Has severe hypersensitivity and adverse events (≥Grade 3) to nivolumab and/or any PD-1/PD-L1 inhibitors.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response | 2 months
  Viable tumor comprised ≤ 10% of resected tumor specimens

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 months
  Partial response is defined as a decrease by 30% or more in sums of longest diameter of measurable target lesions
Positron Emission Tomography (PET)-CT response | 2 months
  Complete metabolic response is defined as the SUV of 2.5 or less than 2.5 of primary tumor
Progression-free survival (PFS) | 24 months
  Time from the enrollment to disease relapse after complete resection or death from any cause
Overall survival (OS) | 24 months
  Time from the enrollment to death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Mu Sun, Principal Investigator — Samsung Medical Center
Locations (1):
- Jong-Mu Sun, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No